CLINICAL TRIAL: NCT07010419
Title: A Global Phase 3, Double-Blind, Randomized, Controlled Multicenter Study to Assess the Efficacy and Safety of Firmonertinib Versus Placebo for Adjuvant Treatment in Participants With Stage IB - IIIB NSCLC With Uncommon Epidermal Growth Factor Receptor (EGFR) Mutations, Following Complete Surgical Resection With or Without Adjuvant Chemotherapy (FIRMOST)
Brief Title: A Study to Assess the Efficacy and Safety of Firmonertinib Versus Placebo for Adjuvant Treatment in Participants With Stage IB - IIIB NSCLC With Uncommon Epidermal Growth Factor Receptor (EGFR) Mutations, Following Complete Surgical Resection With or Without Adjuvant Chemotherapy（FIRMOST）
Acronym: FIRMOST
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Collaborators: ArriVent BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FURMO-005
Record Dates: First submitted 2025-05-20; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: NSCLC; Adjuvant Treatment
Keywords: EGFR; NSCLC; Firmonertinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Firmonertinib (Experimental): Firmonertinib: 240 mg, QD, orally
  Interventions: Drug: Firmonertinib
- Placebo (Placebo Comparator): Placebo: 240 mg, QD, orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Firmonertinib — Firmonertinib: 240 mg, QD, orally
  Arms: Firmonertinib
Drug: Placebo — Placebo: 240 mg, QD, orally
  Arms: Placebo

SUMMARY:
This is a Phase 3, global, double-blind, randomized, controlled multicenter clinical study to assess the efficacy and safety of adjuvant treatment with firmonertinib versus placebo in participants with Stage IB-IIIB NSCLC with uncommon EGFR mutations (exon 20 insertions, PACC and classical-like mutations) after complete surgical resection with or without adjuvant chemotherapy.

About 338 eligible participants will be enrolled and randomized in a 1:1 ratio to receive either firmonertinib 240 mg QD or placebo QD in 21-day treatment cycles. Before randomization, the participant must have undergone complete surgical resection (R0 resection), must have sufficiently recovered from surgery, and must have completed adjuvant chemotherapy (if applicable). The participants will receive firmonertinib or placebo as adjuvant treatment until unacceptable toxicity, withdrawal of informed consent, disease recurrence, initiation of new antitumor treatment, completion of treatment, or other end of treatment reason is met.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the Informed Consent Form (ICF).
2. Aged ≥ 18 years old. Participants from Japan/Taiwan aged ≥ 20 years old.
3. Histologically confirmed diagnosis of primary non-small cell lung cancer (NSCLC) of predominantly non-squamous histology.
4. Underwent complete surgical resection of primary lung cancer and systematic lymph node dissection (R0 resection).
5. Classified post-operatively as Stage IB, II, IIIA, or IIIB (T3N2M0 only) on the basis of pathologic criteria, with the disease staging following the 9th Edition TNM Staging Classification: Lung Cancer issued by Union for International Cancer Control (UICC) and American Joint Committee on Cancer (AJCC).
6. Documented results of the presence of uncommon EGFR mutations (exon 20 insertion mutations, PACC mutations, and/or classical-like mutations, either as single mutations or as co-mutations), in tumor tissue or blood via a validated NGS or validated PCR assay.

Exclusion Criteria:

A participant would be excluded from the study if he/she meets any of the following:

1. NSCLC with EGFR Exon 19 deletion or L858R or C797S mutation.
2. Incomplete resection (R1/R2) or segmentectomy or wedge resection only.
3. Prior treatment with any of the following:

   1. Prior treatment with any antineoplastic therapy other than standard platinum-based doublet adjuvant chemotherapy.
   2. prior treatment with neoadjuvant therapy.
4. Concurrent malignant tumors other than the primary tumor; participants with cancers that can be treated locally and cured may be eligible.
5. Previous ILD (including drug-induced ILD) or active ILD/active radiation pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2032-04-30 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | Up to 3 years
  DFS as assessed by the investigator in Stage II- IIIB. DFS defined as the time from the date of randomization to the first observation of disease recurrence (by pathological diagnosis or imaging) or death caused by any reason, whichever occurs first.

SECONDARY OUTCOMES:
Disease free survival (DFS) | Up to 3 years
  DFS as assessed by the blinded independent central review (BICR) in Stage II-IIIB
Disease free survival (DFS) | Up to 3 years
  DFS as assessed by the investigator in Stage IB-IIIB; DFS as assessed by the BICR in Stage IB-IIIB
Disease free survival rates | Up to 5 years
  2-, 3-, and 5-year DFS rates as assessed by the investigator and BICR in Stage II-IIIB and in Stage IB-IIIB
Overall survival (OS) | Up to 5 years
  OS defined as the time from the date of randomization to the date of death due to any cause, in Stage II-IIIB and in Stage IB-IIIB
Overall survival rates | Up to 5 years
  2-, 3-, and 5-year OS rates in Stage II-IIIB and in Stage IB-IIIB
Adverse event (AE) | Up to 5 years
  Incidence and severity of AEs, with severity as determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Master, Principal Investigator — Sun Yat-sen University; Fan Yang, Doctor, Principal Investigator — Peking University People's Hospital
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangdong, Guangzhou